CLINICAL TRIAL: NCT03374488
Title: A Phase 3 Randomized, Double-Blind Clinical Study of Pembrolizumab + Epacadostat vs Pembrolizumab + Placebo as a Treatment for Recurrent or Progressive Metastatic Urothelial Carcinoma in Patients Who Have Failed a First-Line Platinum-containing Chemotherapy Regimen for Advanced/Metastatic Disease (KEYNOTE-698/ECHO-303)
Brief Title: Pembrolizumab + Epacadostat vs Pembrolizumab + Placebo in Recurrent or Progressive Metastatic Urothelial Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KEYNOTE-698/ECHO-303; 2017-002310-31 (EudraCT Number)
Record Dates: First submitted 2017-12-11; First posted 2017-12-15 (Actual); Results first posted 2019-08-28 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: UC (Urothelial Cancer)
Keywords: Urothelial carcinoma; programmed cell death protein 1 (PD-1) inhibitor; indoleamine 2,3-dioxygenase (IDO) inhibitor
MeSH Terms: conditions — Carcinoma, Transitional Cell; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; epacadostat

STUDY DESIGN:
Masking Description: The study will be unblinded after the last participant completes Week 9 imaging assessment for efficacy analysis and after appropriate EC/IRB approvals have been received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab 200 mg + Epacadostat 100 mg BID (Experimental): Pembrolizumab + epacadostat
  Interventions: Drug: Pembrolizumab; Drug: Epacadostat
- Pembrolizumab 200 mg + placebo BID (Active Comparator): Pembrolizumab + placebo
  Interventions: Drug: Pembrolizumab; Drug: Placebo

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab administered intravenously Day 1 of each cycle every 3 weeks.
  Other Names: MK-3475
Drug: Epacadostat — Epacadostat administered orally twice daily.
  Other Names: INCB024360
  Arms: Pembrolizumab 200 mg + Epacadostat 100 mg BID
Drug: Placebo — Matching placebo administered orally twice daily.
  Arms: Pembrolizumab 200 mg + placebo BID

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of pembrolizumab + epacadostat vs pembrolizumab + placebo as a treatment for recurrent or progressive metastatic urothelial carcinoma in patients who have failed a first-line platinum-containing chemotherapy regimen for advanced/metastatic disease.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed diagnosis of urothelial carcinoma of the renal pelvis, ureter, bladder, or urethra, that is transitional cell, or mixed transitional/non-transitional (predominantly transitional) cell type.
* Progression or recurrence of urothelial carcinoma following one prior platinum containing chemotherapy regimen for metastatic or unresectable locally advanced disease. A participant who receives a neoadjuvant or adjuvant platinum-containing regimen following cystectomy for localized muscle-invasive urothelial carcinoma is acceptable (without further systemic treatment), if recurrence/progression occurs ≤ 12 months following completion of therapy.
* Measurable disease based on RECIST v1.1.
* Have provided an archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated for PD-L1 analysis.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate organ function per protocol-defined criteria.

Exclusion Criteria:

* Urothelial carcinoma that is suitable for local therapy with curative intent.
* History or presence of an abnormal electrocardiogram (ECG) that, in the investigator's opinion, is clinically meaningful.
* Known additional malignancy that is progressing or has required active treatment within the past 3 years.
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, ie, without evidence of progression for at least 4 weeks by repeat imaging.
* Active autoimmune disease that has required systemic treatment in past 2 years.
* Known history of human immunodeficiency virus (HIV) infection. HIV testing is not required unless mandated by local health authority.
* Known history of or is positive for active hepatitis B (HBsAg reactive) or has active hepatitis C (HCV RNA). Note: Testing must be performed to determine eligibility.
* Use of protocol-defined prior/concomitant therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-12-22 (Actual); Primary Completion 2018-07-27 (Actual); Study Completion 2020-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Jones, MD, Study Director — Incyte Corporation
Locations (135):
- United States (24):
  - Ironwood Cancer & Research Centers, Chandler, Arizona
  - University of California Irvine Medical Center, Orange, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - UCLA Hematology Oncology Santa Monica, Santa Monica, California
  - Smilow Cancer Center at Yale-New Haven, New Haven, Connecticut
  - Northside Hospital, Inc. - GCS/Annex, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Quincy Medical Group, Quincy, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - NYU Clinical Cancer Center, New York, New York
  - Oklahoma Cancer Specialists & Research Institute, Tulsa, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina-Hollings Cancer Center, Charleston, South Carolina
  - University of Tennessee Medical Center Knoxville, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - US Oncology and Research, Fort Worth, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - VCU Massey Cancer Center, Richmond, Virginia
- Australia (4):
  - Southern Medical Day Care Centre, Wollongong, New South Wales
  - Austin Health-Austin Hospital, Heidelberg, Victoria
  - Adelaide Cancer Centre, Kurralta Park
  - Macquarie University Hospital, Macquarie Park
- Canada (6):
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - CIUSSS - Hopital Maisonneuve- Rosemont, Montreal, Quebec
  - CIUSSS de l Est de L Ile de Montreal - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - CHU de Quebec-Universite Laval-Hotel Dieu de Quebec, Québec, Quebec
- Denmark (4):
  - Aalborg University Hospital, Aalborg
  - Rigshospitalet, Copenhagen
  - Herlev Hospital, Herlev
  - Sjaellands Universitetshospital Naestved, Næstved
- France (13):
  - Institut de Cancerologie de l Ouest Site Paul Papin, Angers
  - Clinique Sainte Catherine, Avignon
  - Centre de Lutte Contre le Cancer Francois Baclesse, Caen
  - Clinique Victor Hugo, Le Mans
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Institut du Cancer de Montpellier, Montpellier
  - Hopital Cochin, Paris
  - Hopital Saint Louis, Paris
  - Institut Jean Godinot, Reims
  - Centre Medico-Chirurgical Foch, Suresnes
  - C.H.U. de Tours - Hopital Bretonneau, Tours
  - Institut Gustave Roussy, Villejuif
- Germany (7):
  - Universitaetsklinikum Schleswig-Holstein. Campus Luebeck, Lübeck, Schleswig-Holstein
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - Universitatsklinikum Hamburg-Eppendorf, Hamburg
  - Universitaetsklinikum Jena, Jena
  - Universitaetsklinikum Magdeburg A.o.R., Magdeburg
  - Klinikum rechts der Isar der Technischen Universitat, München
  - Universitaetsklinikum Tuebingen, Tübingen
- Hungary (6):
  - Orszagos Onkologiai Intezet, Budapest
  - Uzsoki Utcai Korhaz, Budapest
  - Somogy Megyei Kaposi Mor Oktato Korhaz, Kaposvár
  - Borsod-Abauj-Zemplen Megyei Korhaz es Egyetemi Oktato Korhaz, Miskolc
  - Pecsi Tudomanyegyetem AOK, Pécs
  - Jasz - Nagykun Szolnok megyei Hetenyi Geza Korhaz - Rendelointezet, Szolnok
- Ireland (6):
  - Cork University Hospital, Cork
  - Beaumont Hospital, Dublin
  - Adelaide & Meath Hospital (Incl NCH), Dublin
  - University College Hospital Galway, Galway
  - University Hospital Limerick, Limerick
  - Waterford Regional Hospital, Waterford
- Israel (7):
  - Soroka Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Sourasky Medical Center, Tel Aviv
  - Assaf Harofeh Medical Center, Ẕerifin
- Italy (5):
  - Medical Oncology Ospedale San Donato, Arezzo
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Istituto Nazionale Tumori Fondazione Pascale, Napoli
  - Istituto Oncologico Veneto, Padua
- Japan (8):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - Nara Medical University Hospital, Kashihara, Nara
  - Yamaguchi University Hospital, Ube, Yamaguchi
  - Osaka International Cancer Institute, Osaka
  - Medical Hospital, Tokyo Medical And Dental University, Tokyo
  - Yusen Logistics Co Ltd,. Haneda Logistics Center (MSD DC), Tokyo
- Netherlands (5):
  - Antoni van Leeuwenhoek Ziekenhuis, Amsterdam
  - VU University Medical Center, Amsterdam
  - Amphia Ziekenhuis, Breda
  - Catharina Ziekenhuis, Eindhoven
  - University Medical Center Groningen, Groningen
- Russia (8):
  - Leningrad Regional Oncology Dispensary, Saint Petersburg, Leningrad Region, Vsevolozhsky District
  - Ivanovo Regional Oncology Dispensary, Ivanovo
  - N.N. Blokhin NMRCO, Moscow
  - Russian Scientific Center of Roentgenoradiology, Moscow
  - National Medical Research Radiological Centre, Moscow
  - Ryazan Regional Clinical Oncology Dispensary, Ryazan
  - Pokrovskaya City Hospital, Saint Petersburg
  - Clinic of Bashkortostan State Medical University, Ufa
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (8):
  - Hospital del Mar, Barcelona
  - Hospital Vall D Hebron, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - MD Anderson Cancer Center Madrid, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela
  - Instituto Valenciano de Oncologia, Valencia
- Taiwan (5):
  - Chang Gung Medical Foundation. Kaohsiung Branch, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Turkey (Türkiye) (8):
  - Adana Sehir Hastanesi, Adana
  - Dr. Abdurrahman Yurtaslan Ankara Onkoloji EAH, Ankara
  - Akdeniz Universitesi Tip Fakultesi, Antalya
  - Pamukkale Unv. Tip Fak., Denizli
  - Trakya Universitesi Tip Fakultesi, Edirne
  - Marmara Universitesi Pendik Arastirma ve Uyg. Hastanesi, Istanbul
  - Dokuz Eylul University Faculty of Medicine, Izmir
  - Samsun Medical Park Hastanesi, Samsun
- United Kingdom (7):
  - Royal Marsden NHS Trust, Sutton, Surrey
  - Queen Elizabeth Hospital, Birmingham
  - Barts Health NHS Trust - St Bartholomew s Hospital, London
  - Royal Free London NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - Plymouth Hospitals NHS Trust, Plymouth
  - Sunderland Royal Hospital, Sunderland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cicin I, Plimack ER, Gurney H, Leibowitz R, Alekseev BY, Parnis FX, Peer A, Necchi A, Bellmunt J, Nishiyama H, Clark J, Munteanu M, Kataria R, Jia C, Powles T, Sternberg CN. Epacadostat plus pembrolizumab versus placebo plus pembrolizumab for advanced urothelial carcinoma: results from the randomized phase III ECHO-303/KEYNOTE-698 study. BMC Cancer. 2024 Jul 25;23(Suppl 1):1256. doi: 10.1186/s12885-023-11213-6. PMID 39054485

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 82 centers in 16 countries.
Groups:
- Pembrolizumab 200 mg + Epacadostat 100 mg BID: Pembrolizumab administered intravenously Day 1 of each cycle every 3 weeks. Epacadostat administered orally twice daily.
- Pembrolizumab 200 mg + Placebo BID: Pembrolizumab administered intravenously Day 1 of each cycle every 3 weeks. Matching placebo administered orally twice daily.
Period: Overall Study
Arm/Group | Pembrolizumab 200 mg + Epacadostat 100 mg BID | Pembrolizumab 200 mg + Placebo BID
Started | 42 | 42
Intention-to-Treat (ITT) | 42 | 42
All Participants as Treated (APaT) | 42 | 41
Completed (Refers to participants that discontinued study with amendment 4, and didn't require follow-up.) | 23 | 28
Not Completed | 19 | 14
Not completed — Death | 13 | 13
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Physician Decision | 3 | 0

BASELINE CHARACTERISTICS:
Population: The Intention-to-Treat (ITT) population consisted of all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab 200 mg + Epacadostat 100 mg BID | Pembrolizumab 200 mg + Placebo BID | Total
Number analyzed (Participants) | 42 | 42 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (8.7) | 65.2 (10.0) | 66.5 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 35 | 37 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 38 | 37 | 75
  Unknown or Not Reported | 4 | 5 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 5 | 6 | 11
  White | 35 | 32 | 67
  Missing | 2 | 4 | 6
Metastasis Status at Screening [Count of Participants; unit: Participants]
  Metastatic | 35 | 40 | 75
  Advanced/Unresectable | 7 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) With Pembrolizumab + Epacadostat Versus Pembrolizumab + Placebo
Description: ORR was defined as the percentage of participants who had a complete response (CR), disappearance of all target lesions or partial response (PR), >=30% decrease in the sum of the longest diameter of target lesions per RECIST v1.1 by investigator determination.
Time Frame: up to 9 weeks +14 days
Population: The Intention-to-Treat (ITT) population consisted of all randomized participants. Responses are based on Investigator assessments per RECIST 1.1 without confirmation using all scans up to week 9 (day 63) + 14 days.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pembrolizumab 200 mg + Epacadostat 100 mg BID | Pembrolizumab 200 mg + Placebo BID
Number analyzed (Participants) | 42 | 42
percentage of participants | 21.4 [12.49 to 43.26] | 9.5 [3.11 to 26.06]

2. Secondary Outcome: Safety and Tolerability of Pembrolizumab + Epacadostat Versus Pembrolizumab + Placebo as Measured by Number of Participants Experiencing Adverse Events (AEs)
Description: AE is defined as any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Time Frame: Up to 8 months
Population: All Participants as Treated (APaT) population consisted of all randomized participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab 200 mg + Epacadostat 100 mg BID | Pembrolizumab 200 mg + Placebo BID
Number analyzed (Participants) | 42 | 41
Participants | 42 | 39

3. Secondary Outcome: Safety and Tolerability of Pembrolizumab + Epacadostat Versus Pembrolizumab + Placebo as Measured by Number of Participants Discontinuing Study Treatment Due to AE
Description: as for outcome 2
Time Frame: Up to 8 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab 200 mg + Epacadostat 100 mg BID | Pembrolizumab 200 mg + Placebo BID
Number analyzed (Participants) | 42 | 41
Participants | 4 | 6

ADVERSE EVENTS:
Time Frame: Up to 8 months
Groups:
- MK-3475 200 mg Q3W + Epacad: MK-3475 200 mg Q3W + epacad
- MK-3475 200 mg Q3W + Placeb: MK-3475 200 mg Q3W + placeb
- Total: Total
Arm/Group | MK-3475 200 mg Q3W + Epacad | MK-3475 200 mg Q3W + Placeb | Total
All-Cause Mortality (participants affected / at risk) | 14/42 | 18/41 | 32/83
Serious Adverse Events (participants affected / at risk) | 22/42 | 16/41 | 38/83
Other Adverse Events (participants affected / at risk) | 39/42 | 35/41 | 74/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-3475 200 mg Q3W + Epacad (N=42) | MK-3475 200 mg Q3W + Placeb (N=41) | Total (N=83)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Amylase increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (2)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Disease progression (General disorders) | 1 (1) | 0 (0) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2) | 1 (1) | 3 (3)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (10) | 6 (6) | 15 (16)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (5) | 3 (5) | 6 (10)
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-3475 200 mg Q3W + Epacad (N=42) | MK-3475 200 mg Q3W + Placeb (N=41) | Total (N=83)
Abdominal pain (Gastrointestinal disorders) | 6 (7) | 2 (2) | 8 (9)
Amylase increased (Investigations) | 4 (4) | 2 (4) | 6 (8)
Anaemia (Blood and lymphatic system disorders) | 11 (15) | 9 (9) | 20 (24)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (3) | 6 (7)
Asthenia (General disorders) | 4 (5) | 7 (10) | 11 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (5) | 8 (9)
Blood alkaline phosphatase increased (Investigations) | 3 (3) | 1 (1) | 4 (4)
Blood creatinine increased (Investigations) | 4 (4) | 3 (3) | 7 (7)
Chest pain (General disorders) | 1 (1) | 4 (4) | 5 (5)
Constipation (Gastrointestinal disorders) | 14 (16) | 6 (6) | 20 (22)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2) | 7 (7)
Decreased appetite (Metabolism and nutrition disorders) | 13 (15) | 6 (6) | 19 (21)
Diarrhoea (Gastrointestinal disorders) | 9 (15) | 4 (5) | 13 (20)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 1 (2) | 4 (5)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 0 (0) | 3 (3)
Dysuria (Renal and urinary disorders) | 4 (4) | 1 (1) | 5 (5)
Fatigue (General disorders) | 13 (13) | 5 (5) | 18 (18)
Groin pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 4 (4)
Haematuria (Renal and urinary disorders) | 8 (9) | 3 (3) | 11 (12)
Headache (Nervous system disorders) | 1 (1) | 4 (4) | 5 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (5) | 0 (0) | 4 (5)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 3 (3)
Hypothyroidism (Endocrine disorders) | 4 (4) | 1 (1) | 5 (5)
Lipase increased (Investigations) | 5 (10) | 2 (4) | 7 (14)
Lymphopenia (Blood and lymphatic system disorders) | 3 (3) | 2 (6) | 5 (9)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (2) | 6 (7)
Nausea (Gastrointestinal disorders) | 10 (12) | 6 (10) | 16 (22)
Oedema peripheral (General disorders) | 3 (3) | 1 (1) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (9) | 4 (7) | 12 (16)
Pyrexia (General disorders) | 7 (7) | 3 (3) | 10 (10)
Rash (Skin and subcutaneous tissue disorders) | 9 (11) | 4 (6) | 13 (17)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 3 (3)
Renal impairment (Renal and urinary disorders) | 4 (4) | 1 (1) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 0 (0) | 3 (4)
Urinary tract infection (Infections and infestations) | 7 (13) | 6 (9) | 13 (22)
Vomiting (Gastrointestinal disorders) | 6 (7) | 4 (7) | 10 (14)
Weight decreased (Investigations) | 4 (4) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/88/NCT03374488/Prot_SAP_000.pdf